CLINICAL TRIAL: NCT06682962
Title: Transcorneal Electrical Stimulation for the Treatment of Visual Field Defects in Patients With Open-Angle Glaucoma - a Monocentric, Randomized, Double-Masked, Sham-Controlled Pilot Study
Brief Title: Transcorneal Electrical Stimulation for the Treatment of Visual Field Defects in Patients With Open-Angle Glaucoma
Acronym: TES-GPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okuvision GmbH (Industry)
Collaborators: Interdisciplinary Center for Clinical Trials, University Medical Center Mainz (Unknown); University Medical Center of the Johannes Gutenberg University Mainz, Department of Ophthalmology (Unknown); Sponsored by the German Federal Ministry of Education and Research (FKZ 13GW0732A) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TES-GPS; CIV-24-02-045997 (Other: EUDAMED)
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma; Pigment Dispersion Glaucoma; Normal Tension Glaucoma
Keywords: TES; TcES; POAG; OkuStim; Okuvision; Glaucoma; Electrical Stimulation
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Exfoliation Syndrome; Low Tension Glaucoma

STUDY DESIGN:
Intervention Model Description: Patients are assigned 1:1 to one of two different groups: Sham group (sham treatment) or TES group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is masked to the treatment group he or she has been assigned to. The determination of the tolerance threshold and the programming of the stimulation parameters on the OkuStim 2 is carried out by unmasked members of the study team as it is impossible to program the OkuStim 2 without knowing the assignment of the patient to the study group. Examinations relating to the primary, secondary or exploratory endpoints are carried out only by masked team members.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham group (Sham Comparator): 0µA to therapy amplitude, ramping up in 30 seconds; directly followed by 0µA stimulation for 30 minutes.
  Stimulation will be performed once per week, for 30 minutes, for 18 months.
  Interventions: Device: Transcorneal electrical stimulation (TES) with the OkuStim 2 System
- TES group (Experimental): 0µA to therapy amplitude, ramping up in 30 seconds; directly followed by stimulation with the therapy amplitude for 30 minutes.
  Stimulation will be performed once per week, for 30 minutes, for 18 months.
  Interventions: Device: Transcorneal electrical stimulation (TES) with the OkuStim 2 System

INTERVENTIONS:
Device: Transcorneal electrical stimulation (TES) with the OkuStim 2 System — Retinal stimulation is achieved through transcorneal current application: using a thread electrode, a weak current (≤ 1mA) is introduced onto the surface of the eye, which spreads through the eye towards the retina.
  Other Names: OkuStim 2 System; OkuStim System; OkuStim

SUMMARY:
Glaucoma is a progressive optic neuropathy with retinal ganglion cell loss which leads to visual field loss. Open-angle glaucoma is the most common form of glaucoma.

The aim of this pilot study is to evaluate the safety and effectiveness of the treatment of visual field defects using transcorneal electrical stimulation (TES) with the OkuStim 2 System in patients with primary open-angle glaucoma, pseudoexfoliation glaucoma, pigment dispersion glaucoma or normal tension glaucoma.

DETAILED DESCRIPTION:
Electrical stimulation therapy with the OkuStim System can help patients with retinitis pigmentosa and other hereditary retinal diseases slow the progression of visual field defects and thus preserve usable vision for longer. Since degenerative processes in the retina also lead to loss of vision in patients with glaucoma, the desired clinical benefit in this group of patients is also to slow down the decline in the visual field.

This is a prospective, single-center, randomized, sham-controlled, double-masked pilot study in a parallel group design. Patients are assigned 1:1 to one of two different groups: Sham group (sham treatment) or TES with maximum tolerated current intensity below the pain threshold (tolerance threshold). Patients are stimulated in one eye (study eye). Since these are patients with progressive visual field defects and the experimental therapy is being compared with a sham treatment, the patients also receive pressure-lowering eye drops ("treatment as usual", "TAU") to ensure the safety of the study participant. Treatment duration is 18 months for each patient, with application of TES once a week for 30min.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the study, the subjects signed and dated informed consent must be submitted before the start of the screening
2. Age ≥ 40 years
3. Primary open-angle glaucoma, pseudoexfoliation glaucoma, pigment dispersion glaucoma or normal tension glaucoma (according to the EGS criteria) in the study eye
4. Current progression in perimetry of at least 1.5 dB per year in the study eye and mean defect (MD) in the study eye between ≥ 6 and ≤ 12 dB (Octopus visual field) or ≤ -6 and ≥ -12 dB (Humphrey visual field) in the screening examination as the mean value of the two visual field examinations carried out as part of the screening (permitted deviation maximum 2 dB)
5. Visual acuity ≥ 0.2 decimal in the study eye (corresponds to a visual acuity of 0.7 logMAR)
6. The patient must master home stimulation after extensive training.
7. Ability of subject to understand the scope, significance and individual consequences of participation in the study
8. Ability of subject to give consent
9. If both eyes meet the inclusion/exclusion criteria, the eye with the higher MD is selected as the study eye. If the MD is the same in both eyes, the eye with the worse visual acuity will be selected as the study eye. If there is no difference between the eyes, the right eye will be selected as the study eye
10. Negative serum or urine pregnancy test at screening in women of childbearing potential. Participants are considered to be of nonchildbearing potential if they are postmenopausal and have not menstruated for at least 12 months prior to screening or if they are surgically sterile
11. Women of childbearing potential must agree to be abstinent or to use highly effective methods of contraception that result in a failure rate of less than 1% per year. This applies consistently throughout the duration of the treatment once you have given your consent to participate in the study.

Exclusion Criteria:

1. Neovascularisations of any origin in the study eye
2. Condition after arterial or venous occlusions in the study eye
3. Condition after intraocular surgery in the last 3 months before the screening examination in the study eye
4. Acute (intra)ocular inflammation in any eye
5. Non-proliferative or proliferative diabetic retinopathy in the study eye
6. Condition after retinal detachment in the study eye
7. Dry age-related macular degeneration affecting the visual field in the study eye
8. Exsudative age-related macular degeneration in the study eye
9. Macular edema of any origin in the study eye
10. Other relevant retinal diseases in the study eye
11. Any form of corneal degeneration that limits vision in the study eye
12. Any disease other than glaucoma affecting the central 30° visual field in the study eye
13. No cataract surgery or other eye surgery may be planned for the patient in the study eye during the duration of the study (except laser trabeculoplasty)
14. Patients with active implants
15. General illnesses that are difficult to control/adjust and which, in the opinion of the investigator, could jeopardize regular study routines
16. Poor general condition according to the investigators assessment
17. Mental illness or dementia, that, in the opinion of the investigator, reduces the understanding of the study procedures and use of the Okustim 2 System
18. Simultaneous participation in another interventional study or past interventions whose effect may still be ongoing (30 days)
19. Breastfeeding women
20. Patients unable to consent
21. Previous enrolment in the TES-GPS study
22. Contraindications to the use of OkuStim 2 such as allergies/hypersensitivity to silver

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Difference in Humphrey visual field examination between the TES-treated group and the sham-treated group | 18 months

SECONDARY OUTCOMES:
Visual field - Changes in the average in the Mean Deviation | 6/12/18 months
Visual field - Changes in local visual field defects in at least 3 positions | 18 months
Visual acuity | 18 months
  Visual acuity measurements will be done using the 4 meter Early Treatment Diabetic Retinopathy Study (ETDRS) protocol.
Intraocular pressure | 18 months
OCT | 18 months
  GCL-OCT (macular cube), thickness
OCT | 18 months
  OCT optic nerve (RNFL), thickness
Flavoprotein fluorescence | 18 months
  Flavoprotein fluorescence (FPF) will be measured with the OcuMet Beacon. FPF will be reported both by intensity (a cumulative value reflecting global signal strength), and heterogeneity (measures variation of the relative intensity across the image).
NEI-VFQ-25 | 18 months
  Original numeric values from the survey are converted to a 0 to 100 scale (scores represent the achieved percentage of the total possible score).
  To calculate an overall composite score for the VFQ-25, the vision-targeted subscale scores are averaged.
Additional antiglaucoma therapies | 18 months
  Comparison between groups regarding additional antiglaucomatous therapies (nature and number of e.g. eye drops, surgery, laser treatments)

OTHER OUTCOMES:
Safety | 18 months
  Safety endpoints are the long-term safety of the device, its tolerability assessed by adverse events and the use of rescue treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Lorenz, Prof., Principal Investigator — Augenklinik und Poliklinik der Universitätsmedizin Mainz, Johannes Gutenberg-Universität Mainz
Locations (1):
- Augenklinik und Poliklinik der Universitätsmedizin Mainz, Johannes Gutenberg-Universität Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenz K, Schuster A, Michel HM, Ruckes C, Kronfeld K, Schippert R, Stett A, Beck A. Transcorneal electrical stimulation for the treatment of visual field defects in patients with open-angle glaucoma: a monocentric, randomised, double-masked, sham-controlled pilot study: the TES-GPS study protocol. BMJ Open. 2026 Feb 9;16(2):e112879. doi: 10.1136/bmjopen-2025-112879. PMID 41663170